CLINICAL TRIAL: NCT04955301
Title: Can we Prime Sustainable Food Choice? A Mix-methods Study
Brief Title: Consumers' Preference for Sustainable Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Qiuyan Liao, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201901231sv_a
Record Dates: First submitted 2021-06-04; First posted 2021-07-08 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Food Consumption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control message group (No Intervention): Participants will not receive the priming manipulation.
- Health benefits priming group (Experimental): Participants will be cueing with health benefits by asking to do a word-search exercise beginning with: "In the following, please choose words/statements that can indicate that having a healthy and sustainable diet can have health benefits, such as..."
  Interventions: Behavioral: Priming intervention
- Environmental benefits priming group (Experimental): Participants will be cueing with environmental benefits by asking to do a word-search exercise beginning with: "In the following, please choose words/statements that can indicate that having a healthy and sustainable diet can have environmental benefits, such as..."
  Interventions: Behavioral: Priming intervention
- Environmental and health co-benefits priming group (Experimental): Participants will be cueing with environmental and health co-benefits by asking to do a word-search exercise beginning with: "In the following, please choose words/statements that can indicate that having a healthy and sustainable diet can have both benefits for health and the environment, such as..."
  Interventions: Behavioral: Priming intervention

INTERVENTIONS:
Behavioral: Priming intervention — The priming manipulation will be embedded in one discrete choice experiment to test the effect of three priming interventions: priming with health benefits, environment benefits, and co-benefits of having sustainable diets, respectively, on consumers' preference for sustainable foods, and the relative importance of proximal attributes (e.g. taste and price) and distant attributes (e.g., attributes related to environmental sustainability) in determining food choice preference, as well as testing whether the effects of these three priming interventions can be modified by consumers' social orientation values. The cueing manipulation will be achieved by asking participants to complete a word-search exercise.
  Arms: Environmental and health co-benefits priming group; Environmental benefits priming group; Health benefits priming group

SUMMARY:
This study aims to test and compare the effectiveness of three priming interventions on consumers' selection of sustainable foods: priming with environmental benefits, health benefits and co-benefits (environment and health benefits).

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be aged 18 years or above
* Hong Kong residents
* Be able to read Chinese

Exclusion Criteria:

* Subjects who have vegan or vegetarian diets
* Subjects who have to follow special diets due to illnesses will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Consumers' preference for choosing sustainable foods measured by Discrete Choice Experiment | Within 1 day of randomization
  * Measure name: consumers' food consumption preference
  * Measure tool: an online discrete choice experiment
  * Measure units: The frequency of choosing sustainable food

SECONDARY OUTCOMES:
Measure participants' social orientation value using Social Orientation Value Scale | Within 1 day of randomization
  * Measure name: Social Orientation Value (SVO)
  * Measure tool: survey questionnaire
  * Measure units: subjects can slide along a continuum of own-other payoff allocations, measure units should be the times participants choose own or self.

CONTACTS AND LOCATIONS:
Locations (1):
- HKU School of Public Health, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request from PI.